CLINICAL TRIAL: NCT00402623
Title: The Effect of Quercetin on the Increased Inflammatory and Decreased Antioxidant Status in Sarcoidosis
Brief Title: The Effect of Quercetin in Sarcoidosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Dr. A.W. Boots, Maastricht University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MEC 05.142.5
Record Dates: First submitted 2006-11-20; First posted 2006-11-22 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2008-02

CONDITIONS: Sarcoidosis
Keywords: sarcoidosis; quercetin; supplementation; oxidative stress; inflammation
MeSH Terms: conditions — Sarcoidosis; Inflammation | interventions — Quercetin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): placebo
  Interventions: Other: placebo
- 2 (Active Comparator): quercetin (food supplement)
  Interventions: Dietary Supplement: quercetin

INTERVENTIONS:
Dietary Supplement: quercetin — 1000 mg quercetin within 24 hours
  Arms: 2
Other: placebo
  Arms: 1

SUMMARY:
The exact cause of the chronic lung disease sarcoidosis is still unknown. Consequently, a complete efficacious treatment is still not available. Earlier studies indicate an important key role for oxidative stress, i.e. an imbalance between the production of and the protection against ROS, in the etiology of sarcoidosis. Antioxidants, needed for protection against ROS, are indeed lower in sarcoidosis. Therefore, antioxidant therapy to strengthen the reduced antioxidant defense might be efficacious in sarcoidosis treatment. Since ROS are also capable of initiating and mediating inflammation, antioxidant therapy might also mitigate the elevated inflammation that occurs in sarcoidosis. The flavonoid quercetin possesses both anti-oxidative and anti-inflammatory capacities and might therefore serve as a good candidate for antioxidant therapy in sarcoidosis.

Therefore, the aim of the present study is to determine the effect of quercetin supplementation in sarcoidosis patients on markers of both oxidative stress and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of sarcoidosis with emphasize on pulmonary sarcoidosis
* no smoking
* no treatment

Exclusion Criteria:

* clinical diagnosis (and treatment) of other diseases
* symptoms of sarcoidosis in other organs besides the lung
* use of food supplements or vitamins

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-01; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
antioxidant status after 24 hours | 24 hours
inflammatory status after 24 hours | 24 hours

SECONDARY OUTCOMES:
plasma quercetin concentration after 24 hours | 24 hours
plasma malondialdehyde (MDA) levels after 24 hours | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Aalt Bast, PhD, Study Chair — Maastricht University; Agnes W Boots, PhD, Principal Investigator — Maastricht University; Guido R Haenen, PhD, Study Director — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Netherlands

REFERENCES:
- [Derived] Boots AW, Drent M, de Boer VC, Bast A, Haenen GR. Quercetin reduces markers of oxidative stress and inflammation in sarcoidosis. Clin Nutr. 2011 Aug;30(4):506-12. doi: 10.1016/j.clnu.2011.01.010. Epub 2011 Feb 15. PMID 21324570